CLINICAL TRIAL: NCT06086548
Title: Unraveling Metabolic Involvement in Facioscapulohumeral Dystrophy Through Metabolomics
Acronym: METIN-FSHD
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: University of Modena and Reggio Emilia (Other); Federico II University (Other)
Responsible Party: Sponsor
Other Study IDs: 49RC23_0340
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — heparinated plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: patients with molecular diagnosis of facioscapulohumeral dystrophy
  Interventions: Other: metabolomic on plasma sample
- controls: healthy volunteers
  Interventions: Other: metabolomic on plasma sample

INTERVENTIONS:
Other: metabolomic on plasma sample — metabolic phenotyping by plasma metabolomic and mitochondrial biomarker profiling

SUMMARY:
The pathogenesis of facioscapulohumeral dystrophy (FSHD), one of the most prevalent types of inherited muscle disease, is unknown. The reasons underlying its significant clinical heterogeneity, incomplete penetrance, and sex specific differences in the age of onset, are not currently understood. While metabolic changes associated with this disease have so far deserved little attention, recent studies have pinpointed significant metabolic dysregulation as an emerging driving mechanism in the pathophysiology of this untreatable disease. To test this hypothesis, we will perform a deep metabolic phenotyping in a large cohort of highly clinically characterized FSHD patients at different stage of disease and age/sex-matched controls by state-of-art plasma metabolomic and mitochondrial biomarker profiling. These data will allow attributing specific metabolomic signatures to different stages of the disease in each sex. Metabolic pathway analysis will allow gaining insights into the type of metabolic dysregulation associated with the disease pathogenesis, leading to the identification of targeted metabolic/nutritional interventions and biomarker discovery.

ELIGIBILITY:
Inclusion Criteria:

* participant fasting for at least 8 h at the time of blood sampling
* patient with a molecular diagnosis of FSHD (know number of D4Z4 contractions)
* patient with a typical FSHD presentation (at least facial, pelvic ans scapular girdles signs)
* patient with a preserved ability to ambulate at the time of the selection (use of a cane is allowed)

Exclusion Criteria:

* Severe cardiac and respiratory dysfunction.
* Presence of severe systemic diseases unrelated to FSHD.
* Presence of uncontrolled diabetes or hypothyroidism.
* Alcohol or toxic abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruitment of participants will be conducted at Centre Hospitalier Universitaire d'Angers. All subjects will be clinically evaluated on the basis of the CCEF evaluation protocol. Informed consent will be obtained according to the declaration of Helsinki by each participant after explanations on the research protocol and scientific aims.
  Patients will be excluded when they have other disorders that will influence the measurements. Age- and sex-matched healthy subjects will be included through specific calls depending on age.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
metabolic profiling | results should be obtained within 3 months following the inclusion of the last participant
  to perform a detailed metabolic profiling by state-of-art plasma metabolomic coupled to the analysis of GDF15 and FGF21, two recently established biomarkers of mitochondrial dysfunction, in symptomatic FSHD patients of different clinical severity compared to controls

IPD SHARING:
Plan to Share IPD: No